CLINICAL TRIAL: NCT06367374
Title: A Single Arm, Open-label Study of MRD-Guided Zanubrutinib in Combination With Sonrotoclax in Adult Patients With Treatment Naïve Chronic Lymphocytic Leukemia or Small Lymphocytic Lymphoma
Brief Title: MRD Guided Sonrotoclax and Zanubrutinib in Newly Diagnosed CLL/SLL
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Institute of Hematology & Blood Diseases Hospital, China (Other)
Responsible Party: Principal Investigator, Qiu Lugui, Institute of Hematology & Blood Diseases Hospital, China, Institute of Hematology & Blood Diseases Hospital, China
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BGB-11417-2002-IIT；BDH-CLL-004
Record Dates: First submitted 2024-03-20; First posted 2024-04-16 (Actual); Last update posted 2024-04-16 (Actual); Status verified 2024-04

CONDITIONS: Chronic Lymphocytic Leukemia; Small Lymphocytic Lymphoma
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell | interventions — zanubrutinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Sonrotoclax Plus Zanubrutinib (Experimental): * Participants will receive from the start of Cycle 1 a standard dose of zanubrutinib twice daily orally for three cycles and in combination with sonrotoclax starting from Cycle 4 onwards at increasing doses twice a week until the target dose is reached from Cycle 5 and continuing until the end of Cycle 15 (each cycle is 28 days). Patients with a measurable minimal residual disease (MRD) will receive another 12 cycles of Zanubrutinib in combination with sonrotoclax until their MRD is undetectable.
  * Interventions:
    * Drug: Sonrotoclax
    * Drug: Zanubrutinib
  Interventions: Drug: Sonrotoclax; Drug: Zanubrutinib

INTERVENTIONS:
Drug: Sonrotoclax — Participants receive zanubrutinib orally 160mg bid from start of Cycle 1, and in combination with sonrotoclax (SZ) from Cycle 4 onwards at increasing doses until 320mg daily target dose is reached and continuing for at least 12 cycles (each cycle is 28 days).
  Participants with uMRD and PR/CR by the end of Cycle 15 will stop SZ treatment, others will continue to receive SZ for another 12 cycles and stop SZ if uMRD and PR/CR.
  Participants will receive sonrotoclax up to 2 years, and receive zanubrutinib for those with MRD-positive by then.
  Other Names: BGB-11417
Drug: Zanubrutinib — Participants receive zanubrutinib orally 160mg bid from start of Cycle 1,Participants with uMRD and PR/CR by the end of Cycle 15 will stop SZ treatment, others will continue to receive SZ for another 12 cycles and stop SZ if uMRD and PR/CR.
  Participants will receive sonrotoclax up to 2 years, and receive zanubrutinib for those with MRD-positive by then.
  Other Names: BGB- 3111

SUMMARY:
This is a single-arm, open-label study of sonrotoclax plus zanubrutinib with MRD-driven treatment duration in patients with previously untreated Chronic Lymphocytic Leukemia (CLL) or Small Lymphocytic Lymphoma (SLL).

The primary goal of this study is to evaluate the efficacy of MRD-guided zanubrutinib plus sonrotoclax for first-line CLL/SLL treatment.

DETAILED DESCRIPTION:
Chronic lymphocytic leukemia (CLL) and small lymphocytic lymphoma (SLL) are often considered different variations of the same disease due to their many similarities. There is an urgent need for new treatments to improve patients' quality of life, prolong survival, and manage disease-related symptoms.

There are several different methods for treating front-line therapy, including Chemoimmunotherapy (CIT), Bruton tyrosine kinase inhibitors (BTKis), and BCL-2 inhibitors (BCL2is). Continuous treatment with BTK inhibitors is necessary for the treatment of CLL or SLL. However, younger patients may need to limit their therapeutic duration. The combination of BTK inhibitors and BCL-2 inhibitors is believed to be an optimizing regimen that provides a limited duration of therapy.

The main aim of this study is to assess whether MRD-guided zanubrutinib, in combination with sonrotoclax, can be an effective first-line treatment option for adult patients with treatment-naïve CLL or SLL. The goal is to achieve long-lasting and more profound responses, which could allow for the possibility of discontinuing treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Treatment naïve adult patients with diagnosis of CLL/SLL requiring treatment according to iwCLL guidelines 2018
2. Measurable nodal disease by CT/MRI.
3. Adequate hematologic function
4. Adequate hepatic and renal function
5. Eastern Cooperative Oncology Group
6. (ECOG) performance status of 0-2
7. Expected survival period > 6 months

Exclusion Criteria:

1. Any prior systemic therapy used for treatment of CLL/SLL
2. With history of prolymphocytic leukemia, known or currently suspected Richter's transformation
3. Known central nervous system involvement by leukemia or lymphoma
4. Confirmed progressive multifocal leukoencephalopathy (PML)
5. Severe or debilitating pulmonary disease
6. Clinically significant cardiovascular disease
7. Uncontrolled autoimmune hemolytic anemia or idiopathic thrombocytopenia purpura requiring treatment
8. History of other malignancies
9. Prior therapy with study drugs within 4 weeks before screening
10. Active fungal, bacterial, and/or viral infection requiring systemic therapy
11. Known allergy to zanubrutinib or sonrotoclax or any pharmaceutical excipients
12. Pregnant or lactating women
13. Vaccinated with live vaccines within 28 days prior to enrollment
14. Serologically positive of human immunodeficiency virus (HIVAb), or active infection with hepatitis B virus (HBV) or hepatitis C virus (HCV)
15. History of stroke or intracranial hemorrhage within 6 months
16. Requires treatment with a strong cytochrome P450 (CYP) 3A inhibitor

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2024-05-30 (Estimated); Primary Completion 2030-02-28 (Estimated); Study Completion 2030-07-30 (Estimated)

PRIMARY OUTCOMES:
4-Year Progressive Free Survival (PFS) Rate | 4 years after enrollment
  PFS is defined as the time from the date of enrollment to the date of first confirmed disease progression or death due to any cause, whichever occurs first, as determined by investigators

SECONDARY OUTCOMES:
Rate of peripheral blood (PB) and Bone marrow (BM) undetectable minimal residual disease (uMRD) | At screening, the end of Cycle 14 and Cycle 26 (each cycle is 28 days)
  Rate of PB and BM uMRD is defined as proportion of participants achieving remission based on flow cytometry (FCM) result of < 1 CLL cell per 100,000 leukocytes (< 10 ^-4 ), after completion of 12 and 24 cycles of sonrotoclax treatment.
Complete Response Rate (CRR; Complete Response/Complete Response with Incomplete Blood Count Recovery [CR/CRi]) Rate | Up to 4 years
  CR/CRi rate is defined as the percentage of participants achieving a response of complete response (CR), CR with incomplete blood count recovery (CRi) per 2018 IWCLL criteria, as determined by investigators
Overall Response Rate (ORR) | Up to 4 years
  ORR is defined as the percentage of participants achieving a response of complete response (CR), CR with incomplete blood count recovery (CRi), nodular partial response (nPR), partial response (PR), or PR with lymphocytosis (PRL) evaluated under the 2018 IWCLL criteria, as determined byinvestigators
Duration of Response (DOR) | Up to 4 years
  DOR was calculated for participants achieving a response (CR, CRi, nPR, PR) based on 2018 IWCLL response criteria in CLL or a response (PR or better) based on 2014 Lugano response criteria and defined as the interval between the date of initial documentation of a response mentioned above until disease progression (PD) or death from any cause, whichever occurred first
Progression Free Survival (PFS) | Up to 4 years
  PFS is defined as the time from the date of enrollment to the date of first confirmed disease progression or death due to any cause, whichever occurs first, as determined by investigators
Overall Survival (OS) | Up to 4 years
  OS is defined as time from the date of enrollment to the date of death because of any cause
Time to Next Therapy (TTNT) | Up to 4 years
  Time to next CLL or SLL therapy is defined as the time from the first administration of study drugs to the first administration of the next CLL/SLL treatment, as determined by investigators
Overall survival rate | Up to 4 years
  Number, time frame and seriousness of participants with Treatment-Emergent Adverse Events (NCI-TEAE v5.0)

CONTACTS AND LOCATIONS:
Overall Officials: Lugui Qiu, Principal Investigator — Institute of Hematology & Blood Diseases Hospital, China